CLINICAL TRIAL: NCT04334850
Title: Use of a Respiratory Multiplex PCR and Procalcitonin to Reduce Antibiotics Exposure in Patients With Severe Confirmed COVID-19 Pneumonia : a Multicenter, Parallel-group, Open-label, Randomized Controlled Trial
Brief Title: Use of a Respiratory Multiplex PCR and Procalcitonin to Reduce Antibiotics Exposure in Patients With Severe Confirmed COVID-19 Pneumonia
Acronym: MultiCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200392; 2020-001324-33 (EudraCT Number)
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Pneumonia
Keywords: COVID-19 pneumonia; respiratory multiplex PCR; Procalcitonin; Antibiotics saving; Diagnosis; Treatment
MeSH Terms: conditions — COVID-19; Pneumonia; Disease | interventions — Procalcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted antibiotic treatment according to the results of mPCR (Experimental): a broad panel respiratory Mpcr FA-PPP is performed on respiratory tract sample (tracheal aspirate, BAL or sputum), collected 12 hours after inclusion. An algorithm of early antibiotic adaptation and discontinuation, based on the microbiological results, including the mPCR FA-PPP results, and the procalcitonin values and kinetics will be used. This algorithm will be applied as soon as possible after inclusion, and repeated day after day until D7.
  Interventions: Procedure: Combined use of a respiratory broad panel multiplex PCR and procalcitonin
- Control arm (Other): The antimicrobial therapy is left at the discretion of the physicians, as in usual practice.
  Interventions: Other: Usual antibiotic treatment

INTERVENTIONS:
Procedure: Combined use of a respiratory broad panel multiplex PCR and procalcitonin — The actions or procedures added by the research are the application of the algorithm of early antibiotics de-escalation and discontinuation.
  Arms: Targeted antibiotic treatment according to the results of mPCR
Other: Usual antibiotic treatment — The antimicrobial therapy is left at the discretion of the physicians, as in usual practice.
  Arms: Control arm

SUMMARY:
The novel coronavirus SARS-CoV-2 (COVID-19) is an emerging respiratory virus that causes pneumonia. WHO data reported admission to the intensive care unit (ICU) for 6% of patients, with a mortality rate reaching 45%. To date, apart from therapeutic trials, ICU management is symptomatic, based on organ failure support therapies. In the initial phase, the therapeutic management also includes empiric antimicrobial therapy (90% of patients, in accordance with LRTI guidelines (ATS 2019) and SRLF Guidelines (2020). One challenge for the ICU physicians is the timing for discontinuation of antimicrobial treatment, especially in case of shock or ARDS, considering that a substantial proportion of COVID-19 pneumonia patients may have pulmonary bacterial coinfection/superinfection. In order to avoid unnecessary prolonged antimicrobial therapy, and subsequent selective pressure, two tests could be combined in a personalized antibiotic strategy:

* Procalcitonin (PCT): PCT is a useful tool to guide antibiotics discontinuation in community-acquired pneumonia) and viral pneumonia (PMID24612487).
* Respiratory multiplex PCR FA-PPP (Biomérieux®): panel has been enlarged, including 8 viruses and 18 bacteria (quantitative analysis). The turnaround time is short. Sensitivity is high (99%, PMID32179139). It may contribute, in combination with conventional tests, to accelerate and improve the microbiological diagnosis during severe COVID-19 pneumonia.

The hypothesize of the study is that the combination of the mPCR FA-PPP and PCT could be used to reduce antibiotics exposure in patients with severe confirmed COVID-19 pneumonia, with a higher clinical efficacy and safety as compared with a conventional strategy.

DETAILED DESCRIPTION:
Inclusion (D0_H0) is performed in ICU as soon as possible, once the diagnosis of COVID-19 pneumonia is confirmed. Therefore, inclusion might be performed either on ICU admission (if the COVID-19 pneumonia has been confirmed in the pre-ICU wards) or during the ICU stay (if the COVID-19 pneumonia was confirmed after ICU admission). Conventional microbiological investigations are left at the discretion of the physicians, and may include blood cultures, Streptococcus pneumoniae and Legionella pneumophila urinary antigen assays, and a respiratory tract sample for Gram stain examination and 2 days-long culture (if not already done in the past 24 hours). Usual biology includes procalcitonin measurement. Empirical antimicrobial therapy combines a third-generation cephalosporin and a macrolide, or broader-spectrum antibiotics if risk factors for resistant bacteria are identified.

Randomization is performed immediately after the inclusion.

* In the intervention arm, a broad panel respiratory Mpcr FA-PPP is performed on respiratory tract sample (tracheal aspirate, BAL or sputum), collected 12 hours after inclusion. An algorithm of early antibiotic adaptation and discontinuation, based on the microbiological results, including the mPCR FA-PPP results, and the procalcitonin values and kinetics will be used. This algorithm will be applied as soon as possible after inclusion, and repeated day after day until D7.
* In the control arm, the antimicrobial therapy is left at the discretion of the physicians, as in usual practice.

Evaluation criteria are collected at hospital discharge or at D28, and D90. The vital status may be obtained by phone call at D28 (if the patient has been discharged before D28) and at D90.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>= 18 years) admitted to the ICU;
* Severe confirmed COVID-19 pneumonia, defined by i) a newly-appeared pulmonary parenchymal infiltrate; and ii) a positive RT-PCR (either upper or lower respiratory tract) for COVID-19 (SARS-CoV-2); iii) and admission to the ICU or intermediate care unit;
* Informed consent or emergency procedure.

Exclusion Criteria:

* Pregnancy ;
* Congenital immunodeficiency;
* HIV infection with CD4 count below 200/mm3 or unknown in the last year;
* High-grade hematological malignancy;
* Neutropenia (<1 leucocyte/mL or < 0.5 neutrophil/mL);
* Immunosuppressive drugs within the previous 30 days, including anti-cancer cytotoxic chemotherapy and anti-rejection drugs for organ/bone marrow transplant;
* Moribund patient or death expected from underlying disease during the current admission;
* Patient deprived of liberty or under legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Number of antibiotic free days | Day 28
  the number of days alive without any antibiotics at Day 28. The D28 time point is usual in studies assessing antibiotics saving in ICU patients.

SECONDARY OUTCOMES:
Mortality rates | Day 28 and Day 90
Number of defined daily dose (DDD) per 100 patient-days of broad- and narrow-spectrum antibiotics. | day 28
Antibiotics duration at D28 | Day 28
  Total exposure to antibiotics
Number of organ-failure free days (based on SOFA) | Day 28
Incidence rates of bacterial super-infections | day 28
Incidence rates of colonization/infection with multidrug resistant bacteria and Clostridium difficile infections | Day 28
ICU and hospital lengths of stay | Day 28
Quality of life Quality of life | Day 90
  using a quality of life questionnaire (EQ5D5L)

CONTACTS AND LOCATIONS:
Overall Officials: Muriel FARTOUKH, PU-PH MD PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive care department-Hospital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: No